CLINICAL TRIAL: NCT00870740
Title: A Double-Blind, Multicenter, Extension Study to Evaluate the Safety and Efficacy of DAC HYP in Subjects With Multiple Sclerosis Who Have Completed Treatment in Study 205MS201 (SELECT)
Brief Title: Safety and Efficacy Extension Study of Daclizumab High Yield Process (DAC HYP) in Participants With Multiple Sclerosis Who Have Completed Study 205MS201 (NCT00390221) to Treat Relapsing-Remitting Multiple Sclerosis
Acronym: SELECTION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 205-MS-202; EUDRA CT No.: 2008-005559-46
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Results first posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-07

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: MS; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — daclizumab HYP

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1: DAC HYP 150 mg (Experimental): Participants who received placebo in 205MS201 receive DAC HYP 150 mg subcutaneous (SC) injection every 4 weeks for a total of 13 doses.
  Interventions: Biological: BIIB019 (Daclizumab High Yield Process)
- Group 1: DAC HYP 300 mg (Experimental): Participants who received placebo in 205MS201 receive DAC HYP 300 mg SC injection every 4 weeks for a total of 13 doses.
  Interventions: Biological: BIIB019 (Daclizumab High Yield Process)
- Group 2: Washout then DAC HYP 150 mg (Experimental): Participants who received DAC HYP 150 mg SC injection in 205MS201 undergo a washout period (placebo SC every 4 weeks for a total of 5 doses) and then receive DAC HYP 150 mg SC every 4 weeks for a total of 8 doses.
  Interventions: Biological: BIIB019 (Daclizumab High Yield Process); Drug: Placebo
- Group 2: DAC HYP 150 mg (Experimental): Participants who received DAC HYP 150 mg SC injection in 205MS201 receive DAC HYP 150 mg SC every 4 weeks for a total of 13 doses.
  Interventions: Biological: BIIB019 (Daclizumab High Yield Process)
- Group 3: Washout then DAC HYP 300 mg (Experimental): Participants who received DAC HYP 300 mg SC in 205MS201 undergo a washout period (placebo SC every 4 weeks for a total of 5 doses) and then receive DAC HYP 300 mg SC every 4 weeks for a total of 8 doses.
  Interventions: Biological: BIIB019 (Daclizumab High Yield Process); Drug: Placebo
- Group 3: DAC HYP 300 mg (Experimental): Participants who received DAC HYP 300 mg SC in 205MS201 receive DAC HYP 300 mg SC every 4 weeks for a total of 13 doses.
  Interventions: Biological: BIIB019 (Daclizumab High Yield Process)

INTERVENTIONS:
Biological: BIIB019 (Daclizumab High Yield Process) — SC injection
  Other Names: Daclizumab HYP; DAC HYP
Drug: Placebo — Placebo SC injection
  Arms: Group 2: Washout then DAC HYP 150 mg; Group 3: Washout then DAC HYP 300 mg

SUMMARY:
The primary objective of the study was to assess the safety and immunogenicity of extended treatment with DAC HYP. This evaluation included the following major components:

* An assessment of safety and immunogenicity of extended treatment with DAC HYP when administered to MS subjects who had completed 52 weeks of active therapy with DAC HYP in Study 201.
* An assessment of safety and immunogenicity during a 6-month washout period from DAC HYP.
* An assessment of safety and immunogenicity during reinitiation of therapy with DAC HYP after a 6-month washout period.
* An assessment of safety and immunogenicity of DAC HYP when administered to MS subjects who previously received placebo during Study 201.

The secondary objective is to assess the durability of the effect of DAC HYP on multiple sclerosis (MS) disease activity as measured by brain magnetic resonance imaging (MRI) scans and clinical MS relapses.

DETAILED DESCRIPTION:
This study, an extension to Study 205MS201 (NCT00390221), will evaluate the long-term safety, efficacy, and immunogenicity of DAC HYP in MS. In Study 205MS201, study treatment was scheduled to stop at the Week 52 visit. This extension study will provide for the initiation of active therapy with DAC HYP among participants who received placebo during Weeks 0 through 52 in 205MS201. In addition, participants who received active therapy with DAC HYP during Weeks 0 through 52 in Study 205MS201 will continue DAC HYP therapy or resume DAC HYP therapy after a 6-month washout period in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Participated in Study 205MS201 (NCT00390221) for at least 52 weeks and was compliant with the 205MS201 protocol in the opinion of the Investigator.

Key Exclusion Criteria:

* Subjects with any significant change in their medical status from 205MS201 that would preclude administration of DAC HYP, as determined by the Investigator
* Any subject who has permanently discontinued study treatment in Study 205MS201 except subjects who were unblinded during evaluation of an adverse event (AE) and found to be on placebo
* Planned ongoing treatment with any approved or experimental treatment for MS except for the protocol-allowed use of concomitant interferon-beta

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 517 (Actual)
Dates: Start 2009-02; Primary Completion 2012-05 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (58):
- Czechia (6):
  - Research Site, Brno
  - Research Site, Hraddec Kralove
  - Research Site, Olomouc
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Teplice
- Germany (6):
  - Research Site, Bayreuth
  - Research Site, Erlangen
  - Research Site, Marburg
  - Research Site, Osnabrück
  - Research Site, Regensburg
  - Research Site, Rostock
- Hungary (9):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Esztergom
  - Research Site, Győr
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Siófok
  - Research Site, Zalaegerszeg
- India (6):
  - Research Site, Andra-Pradeash
  - Research Site, Bangalore
  - Research Site, Jaipur
  - Research Site, Kolkata
  - Research Site, Mumbai
  - Research Site, Visakhapatnam
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Warsaw
- Russia (11):
  - Research Site, Kazan'
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Smolensk
  - Research Site, Ufa
  - Research Site, Yaroskavl
- Ukraine (8):
  - Research Site, Chernivtsi
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Kharkiv
  - Research Site, Kiev
  - Research Site, Lviv
  - Research Site, Poltava
  - Research Site, Zaporizhzhya
- United Kingdom (5):
  - Research Site, Devon
  - Research Site, London
  - Research Site, Nottingham
  - Research Site, Sheffield
  - Research Site, Stoke-on-Trent

REFERENCES:
- [Derived] Gold R, Stefoski D, Selmaj K, Havrdova E, Hurst C, Holman J, Tornesi B, Akella S, McCroskery P. Pregnancy Experience: Nonclinical Studies and Pregnancy Outcomes in the Daclizumab Clinical Study Program. Neurol Ther. 2016 Dec;5(2):169-182. doi: 10.1007/s40120-016-0048-2. Epub 2016 Jul 13. PMID 27411694
- [Derived] Giovannoni G, Gold R, Selmaj K, Havrdova E, Montalban X, Radue EW, Stefoski D, McNeill M, Amaravadi L, Sweetser M, Elkins J, O'Neill G; SELECTION Study Investigators. Daclizumab high-yield process in relapsing-remitting multiple sclerosis (SELECTION): a multicentre, randomised, double-blind extension trial. Lancet Neurol. 2014 May;13(5):472-81. doi: 10.1016/S1474-4422(14)70039-0. Epub 2014 Mar 19. PMID 24656609
- See also: The website of the National Multiple Sclerosis Society, an organization dedicated to providing information to individuals with MS, their families and healthcare providers. — http://www.nationalmssociety.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo + DAC HYP 150 mg: Participants who previously received placebo in study 205MS201 (NCT00390221) received DAC HYP 150 mg subcutaneous (SC) injection every 4 weeks for a total of 13 doses.
- Placebo + DAC HYP 300 mg: Participants who previously received placebo in study 205MS201 received DAC HYP 300 mg SC injection every 4 weeks for a total of 13 doses.
- DAC HYP 150 mg + Washout: Participants who previously received DAC HYP 150 mg SC injection in study 205MS201 underwent a washout period (placebo SC every 4 weeks for a total of 5 doses) and then received DAC HYP 150 mg SC every 4 weeks for a total of 8 doses.
- DAC HYP 150 mg for 2 Years: Participants who previously received DAC HYP 150 mg SC injection in study 205MS201 received DAC HYP 150 mg SC every 4 weeks for a total of 13 doses.
- DAC HYP 300 mg + Washout: Participants who previously received DAC HYP 300 mg SC in study 205MS201 underwent a washout period (placebo SC every 4 weeks for a total of 5 doses) and then received DAC HYP 300 mg SC every 4 weeks for a total of 8 doses.
- DAC HYP 300 mg for 2 Years: Participants who previously received DAC HYP 300 mg SC in study 205MS201 received DAC HYP 300 mg SC every 4 weeks for a total of 13 doses.
Period: Overall Study
Arm/Group | Placebo + DAC HYP 150 mg | Placebo + DAC HYP 300 mg | DAC HYP 150 mg + Washout | DAC HYP 150 mg for 2 Years | DAC HYP 300 mg + Washout | DAC HYP 300 mg for 2 Years
Started | 86 (number randomized and dosed) | 84 (number randomized and dosed) | 86 (number randomized and dosed) | 86 (number randomized and dosed) | 88 (number randomized and dosed) | 87 (number randomized and dosed)
Completed | 74 | 75 | 76 | 74 | 77 | 70
Not Completed | 12 | 9 | 10 | 12 | 11 | 17
Not completed — Adverse Event | 2 | 1 | 3 | 2 | 1 | 6
Not completed — Consent Withdrawn | 6 | 3 | 4 | 6 | 6 | 5
Not completed — Investigator Decision | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Subject Non-compliance | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 2 | 5 | 2 | 4 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + DAC HYP 150 mg | Placebo + DAC HYP 300 mg | DAC HYP 150 mg + Washout | DAC HYP 150 mg for 2 Years | DAC HYP 300 mg + Washout | DAC HYP 300 mg for 2 Years | Total
Number analyzed (Participants) | 86 | 84 | 86 | 86 | 88 | 87 | 517
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (9.78) | 37.8 (7.98) | 36.8 (8.76) | 36.2 (9.30) | 36.2 (9.03) | 36.0 (7.60) | 36.9 (8.77)
Age, Customized [Number; unit: participants]
  18 to 19 years | 0 | 0 | 0 | 0 | 1 | 1 | 2
  20 to 29 years | 19 | 13 | 19 | 25 | 20 | 16 | 112
  30 to 39 years | 26 | 37 | 29 | 28 | 35 | 41 | 196
  40 to 49 years | 29 | 28 | 33 | 27 | 24 | 25 | 166
  50 to 55 years | 11 | 6 | 5 | 6 | 7 | 3 | 38
  > 55 years | 1 | 0 | 0 | 0 | 1 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 54 | 59 | 53 | 59 | 48 | 326
  Male | 33 | 30 | 27 | 33 | 29 | 39 | 191

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs)
Description: Treatment-emergent AE: any untoward medical occurrence after the first dose of study treatment that did not necessarily have a causal relationship with this treatment. Serious AE (SAE): any untoward medical occurrence that at any dose: resulted in death; in the view of the Investigator, placed the subject at immediate risk of death (a life-threatening event); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in a congenital anomaly/birth defect. An SAE could also have been a medically significant event that, in the opinion of the Investigator, jeopardized the subject or required intervention to prevent one of the other outcomes listed in the definition above.
Time Frame: Up to 72 weeks
Population: Safety population: all randomized participants who received study treatment. Participants who discontinued study treatment due to an AE and/or withdrew from the study due to an AE that started prior to 205MS202 (NCT00870740) and that was treatment-emergent under 205MS201 (NCT00390221) are included in this summary.
Measure: Number; unit: participants
Arm/Group | Placebo + DAC HYP 150 mg | Placebo + DAC HYP 300 mg | DAC HYP 150 mg + Washout | DAC HYP 150 mg for 2 Years | DAC HYP 300 mg + Washout | DAC HYP 300 mg for 2 Years
Number analyzed (Participants) | 86 | 84 | 86 | 86 | 88 | 87
participants
  Participants with an AE | 61 | 57 | 70 | 57 | 61 | 62
  Participants with a moderate or severe AE | 37 | 33 | 45 | 41 | 35 | 35
  Participants with a severe AE | 1 | 3 | 3 | 2 | 4 | 4
  Participants with a possibly/definitely related AE | 18 | 12 | 24 | 13 | 22 | 22
  Participants with an SAE | 15 | 11 | 18 | 15 | 15 | 11

2. Primary Outcome: Number of Participants With Abnormalities in Vital Signs
Description: For participants who took DAC HYP during 205MS201 (NCT00390221) the baseline is defined as the baseline from 205MS201, and for participants who took placebo during 205MS201 the baseline is defined as the baseline from 205MS202 (NCT00870740). All post-baseline data are taken after first dose in 205MS202 only. SBP=systolic blood pressure; DBP=diastolic blood pressure; bpm=beats per minute; ↑ BL=increase from baseline; ↓ BL=decrease from baseline.
Time Frame: Up to Week 72
Population: Safety population: all randomized participants who received study treatment; n=number of subjects who had a baseline assessment and at least one post-baseline assessment for that vital sign.
Measure: Number; unit: participants
Arm/Group | Placebo + DAC HYP 150 mg | Placebo + DAC HYP 300 mg | DAC HYP 150 mg + Washout | DAC HYP 150 mg for 2 Years | DAC HYP 300 mg + Washout | DAC HYP 300 mg for 2 Years
Number analyzed (Participants) | 86 | 84 | 86 | 86 | 88 | 87
participants
  SBP >180 mmHg w/>40 mmHg ↑ BL; n=86,84,85,85,88,87 | 0 | 0 | 0 | 0 | 0 | 0
  SBP <90 mmHg w/>30 mmHg ↓ BL; n=86,84,85,85,88,87 | 1 | 1 | 0 | 0 | 1 | 0
  DBP >120 mmHg w/>20 mmHg ↑ BL; n=86,84,85,85,88,87 | 0 | 0 | 0 | 0 | 0 | 0
  DBP <50 mmHg w/>20 mmHg ↓ BL; n=86,84,85,85,88,87 | 1 | 0 | 0 | 0 | 0 | 0
  Pulse >120 bpm w/>20 bpm ↑ BL; n=86,84,85,85,88,87 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse <50 bpm w/>20 bpm ↓ BL; n=86,84,85,85,88,87 | 0 | 1 | 1 | 1 | 1 | 0
  Temperature >38C w/≥1C ↑ BL; n=86,84,85,84,88,87 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Adjusted Annualized Relapse Rate
Description: Relapses are defined as new or recurrent neurological symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings upon examination by the Independent Neurology Evaluation Committee (INEC). Relapse rate is calculated as: (Total number of relapses that occurred during the 205MS202 [NCT00870740] treatment phase divided by the total number of days followed in the treatment phase for 205MS202), multiplied by 365 days. Participants who received an alternative multiple sclerosis (MS) medication during 205MS201 (NCT00390221; Year 1) are not included in the summary of relapses and relapse rate for this study (Year 2). Participants are stratified differently in this Outcome Measure as per the pre-specified statistical analysis plan.
Time Frame: Up to 72 weeks
Population: Per-protocol population: all randomized participants who received study treatment, excluding 18 participants from a single site (protocol violation) plus 75 participants for whom the time between the last dose of study treatment in 205MS201 (NCT00390221) and the first dose in 205MS202 (NCT00870740) was 56 days or longer.
Measure: Number (95% Confidence Interval); unit: relapses per person-years
Groups:
- Placebo + DAC HYP: Participants who previously received placebo in study 205MS201 (NCT00390221) received DAC HYP 150 mg or 300 mg SC injection every 4 weeks for a total of 13 doses.
- DAC HYP + Washout: Participants who previously received DAC HYP 150 mg or 300 mg SC injection in study 205MS201 underwent a washout period (placebo SC every 4 weeks for a total of 5 doses) and then received DAC HYP 150 mg or 300 mg SC, respectively, every 4 weeks for a total of 8 doses.
- DAC HYP for 2 Years: Participants who previously received DAC HYP 150 mg or 300 mg SC injection in study 205MS201 received DAC HYP 150 mg or 300 mg SC, respectively, every 4 weeks for a total of 13 doses.
Arm/Group | Placebo + DAC HYP | DAC HYP + Washout | DAC HYP for 2 Years
Number analyzed (Participants) | 163 | 132 | 129
relapses per person-years | 0.179 [0.123 to 0.261] | 0.302 [0.215 to 0.423] | 0.165 [0.105 to 0.259]

4. Secondary Outcome: Estimated Proportion of Participants With a Relapse
Description: Relapses are defined as new or recurrent neurologic symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings upon examination by the INEC. Estimated using Kaplan-Meier analysis where time to first relapse is calculated from date of first dose in the study to date of first confirmed relapse. Participants who received an alternative MS medication before the first relapse were censored at the time of taking the alternative MS medication.
Time Frame: Up to 72 weeks
Population: as for outcome 3
Measure: Number; unit: proportion of participants
Arm/Group | Placebo + DAC HYP 150 mg | Placebo + DAC HYP 300 mg | DAC HYP 150 mg + Washout | DAC HYP 150 mg for 2 Years | DAC HYP 300 mg + Washout | DAC HYP 300 mg for 2 Years
Number analyzed (Participants) | 84 | 79 | 64 | 65 | 68 | 64
proportion of participants | 0.186 | 0.166 | 0.249 | 0.160 | 0.235 | 0.111

5. Secondary Outcome: Mean Number of New Gadolinium-enhancing Lesions
Description: Evaluated by magnetic resonance imaging (MRI) by a central reader. Number of new Gd lesions since the previous scan (the previous scan for Week 20 was Week 52 of study 205MS201 [NCT00390221]). The number of Gd lesions may be imputed using last observation carried forward or using the mean value across all subjects within the treatment group. Baseline visits are not imputed. Participants are stratified differently in this Outcome Measure as per the pre-specified statistical analysis plan.
Time Frame: Week 20, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: lesions
Groups:
- DAC HYP + Washout: Participants who previously received DAC HYP 150 mg or 300 mg SC injection in study 205MS201 (NCT00390221) underwent a washout period (placebo SC every 4 weeks for a total of 5 doses) and then received DAC HYP 150 mg or 300 mg SC every 4 weeks for a total of 8 doses.
- DAC HYP for 2 Years: Participants who previously received DAC HYP 150 mg or 300 mg SC injection in study 205MS201 (NCT00390221) received DAC HYP 150 mg or 300 mg SC every 4 weeks for a total of 13 doses.
Arm/Group | Placebo + DAC HYP | DAC HYP + Washout | DAC HYP for 2 Years
Number analyzed (Participants) | 163 | 132 | 129
lesions
  Week 20 | 0.3 (1.01) | 1.1 (2.34) | 0.2 (0.51)
  Week 52 | 0.2 (0.80) | 0.2 (0.64) | 0.2 (1.21)

6. Secondary Outcome: Mean Number of New or Newly-enlarging T2 Hyperintense Lesions
Description: Lesions detected on T2-weighted sequences represent a range of histopathology related to MS, including edema, inflammation, demyelination, gliosis, and axon loss. Evaluated by MRI by a central reader. New or newly enlarging T2 lesions since baseline of study 205MS202 (NCT00870740). For post-baseline visits, the number of T2 lesions may be imputed using the mean value across all participants within the treatment group, if the participant has non-missing baseline data. Baseline visits are not imputed. Participants are stratified differently in this Outcome Measure as per the pre-specified statistical analysis plan.
Time Frame: Baseline, Week 20, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Placebo + DAC HYP | DAC HYP + Washout | DAC HYP for 2 Years
Number analyzed (Participants) | 156 | 126 | 128
lesions
  Baseline | 46.0 (36.48) | 41.1 (36.36) | 39.8 (32.63)
  Week 20 | 1.1 (2.26) | 2.6 (6.33) | 0.5 (1.28)
  Week 52 | 2.1 (3.68) | 3.3 (6.95) | 1.2 (4.33)

7. Secondary Outcome: Mean Volume of New T1 Hypointense Lesions
Description: T1-weighted scans detect areas of hypointensity that represent a greater degree of tissue destruction and axon loss than T2 hyperintense lesions and are more highly correlated with clinical disability measures and neurological deficit. Evaluated by MRI by a central reader. Baseline is volume of new T1 hypointense lesions since baseline in study 205MS201 (NCT00390221). Scans at Week 20 and Week 52 in 205MS202 are relative to baseline in 205MS202 (NCT00870740). For post-baseline visits, the total volume of T1 lesions may be imputed using the mean value across all subjects within the treatment group. Baseline visits are not imputed.
Time Frame: Baseline, Week 20, Week 52
Population: Per-protocol population: randomized participants who received study treatment, excluding 18 participants from a single site (protocol violation) plus 75 for whom the time between the last dose of study treatment in 205MS201 (NCT00390221) and the first dose in 205MS202 (NCT00870740) was ≥ 56 days; n=participants with measurement at given time point.
Measure: Mean (Standard Deviation); unit: mm^3
Groups:
- Placebo + DAC HYP 300 mg: Participants who previously received placebo in study 205MS201 (NCT00390221) received DAC HYP 300 mg SC injection every 4 weeks for a total of 13 doses.
- DAC HYP 150 mg + Washout: Participants who previously received DAC HYP 150 mg SC injection in study 205MS201 (NCT00390221) underwent a washout period (placebo SC every 4 weeks for a total of 5 doses) and then received DAC HYP 150 mg SC every 4 weeks for a total of 8 doses.
- DAC HYP 150 mg for 2 Years: Participants who previously received DAC HYP 150 mg SC injection in study 205MS201 (NCT00390221) received DAC HYP 150 mg SC every 4 weeks for a total of 13 doses.
- DAC HYP 300 mg + Washout: Participants who previously received DAC HYP 300 mg SC in study 205MS201 (NCT00390221) underwent a washout period (placebo SC every 4 weeks for a total of 5 doses) and then received DAC HYP 300 mg SC every 4 weeks for a total of 8 doses.
- DAC HYP 300 mg for 2 Years: Participants who previously received DAC HYP 300 mg SC in study 205MS201 (NCT00390221) received DAC HYP 300 mg SC every 4 weeks for a total of 13 doses.
Arm/Group | Placebo + DAC HYP 150 mg | Placebo + DAC HYP 300 mg | DAC HYP 150 mg + Washout | DAC HYP 150 mg for 2 Years | DAC HYP 300 mg + Washout | DAC HYP 300 mg for 2 Years
Number analyzed (Participants) | 84 | 79 | 64 | 65 | 68 | 64
mm^3
  Baseline; n=83, 79, 63, 64, 66, 64 | 232.13 (467.811) | 228.90 (390.587) | 126.50 (288.580) | 94.20 (281.450) | 52.26 (184.170) | 44.92 (150.363)
  Week 20; n=81, 74, 62, 65, 63, 63 | 36.17 (114.019) | 62.76 (143.280) | 161.98 (829.086) | 6.29 (24.095) | 12.37 (32.361) | 4.66 (19.386)
  Week 52; n=81, 74, 62, 65, 63, 63 | 88.46 (239.741) | 109.42 (231.734) | 142.31 (628.500) | 17.18 (39.881) | 43.60 (88.084) | 21.42 (82.566)

8. Secondary Outcome: Mean Percentage Change From Baseline in Total Lesion Volume of T2 Hyperintense Lesions
Description: Lesions detected on T2-weighted sequences represent a range of histopathology related to MS, including edema, inflammation, demyelination, gliosis, and axon loss. Evaluated by MRI by a central reader. Baseline values = baseline for study 205MS202 (NCT00870740). For post-baseline visits, the total volume of T2 lesions may be imputed using the mean value across all subjects within the treatment group. Baseline visits are not imputed.
Time Frame: Baseline, Week 52
Population: Per-protocol population (with a baseline and post-baseline assessment): randomized participants who received study treatment, excluding 18 participants from a single site (protocol violation) plus 75 for whom the time between the last dose of study treatment in 205MS201 (NCT00390221) and the first dose in 205MS202 (NCT00870740) was ≥ 56 days.
Measure: Mean (Standard Deviation); unit: percentage change in volume
Arm/Group | Placebo + DAC HYP 150 mg | Placebo + DAC HYP 300 mg | DAC HYP 150 mg + Washout | DAC HYP 150 mg for 2 Years | DAC HYP 300 mg + Washout | DAC HYP 300 mg for 2 Years
Number analyzed (Participants) | 81 | 75 | 62 | 65 | 64 | 63
percentage change in volume | -7.75 (21.952) | -8.44 (13.942) | -0.78 (22.243) | -4.90 (25.935) | -5.40 (16.672) | -8.98 (11.673)

9. Secondary Outcome: Mean Percentage Change From Baseline in Total Volume of Non-gadolinium (Gd)-Enhancing T1 Hypointense Lesions
Description: T1-weighted scans detect areas of hypointensity that represent a greater degree of tissue destruction and axon loss than T2 hyperintense lesions and are more highly correlated with clinical disability measures and neurological deficit. Evaluated by MRI by a central reader. Baseline values = baseline for study 205MS202 (NCT00870740). For post-baseline visits, the total volume of T1 lesions may be imputed using the mean value across all participants within the treatment group. Baseline visits are not imputed.
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage change in volume
Arm/Group | Placebo + DAC HYP 150 mg | Placebo + DAC HYP 300 mg | DAC HYP 150 mg + Washout | DAC HYP 150 mg for 2 Years | DAC HYP 300 mg + Washout | DAC HYP 300 mg for 2 Years
Number analyzed (Participants) | 81 | 74 | 62 | 65 | 63 | 63
percentage change in volume | -3.99 (35.543) | -7.15 (39.932) | -5.51 (49.970) | -13.89 (18.089) | -6.72 (22.721) | -16.59 (17.436)

10. Primary Outcome: Number of Participants With Potentially Clinically Significant Hematology Laboratory Abnormalities
Description: Hematology parameters evaluated include: white blood cells, lymphocytes, neutrophils, red blood cells (RBC), hemoglobin, and platelets.
Time Frame: Up to 72 Weeks
Population: Number of participants in the safety population (all randomized participants who received study treatment) with at least one post-baseline value.
Measure: Number; unit: participants
Arm/Group | Placebo + DAC HYP 150 mg | Placebo + DAC HYP 300 mg | DAC HYP 150 mg + Washout | DAC HYP 150 mg for 2 Years | DAC HYP 300 mg + Washout | DAC HYP 300 mg for 2 Years
Number analyzed (Participants) | 85 | 84 | 85 | 85 | 88 | 87
participants
  White Blood Cell Count <3.0*10^9 cells/L | 0 | 3 | 3 | 4 | 3 | 2
  White Blood Cell Count ≥16.0*10^9 cells/L | 4 | 2 | 1 | 1 | 3 | 1
  Lymphocytes <0.8*10^9 cells/L | 5 | 4 | 6 | 3 | 2 | 5
  Lymphocytes <0.5*10^9 cells/L | 1 | 0 | 1 | 1 | 1 | 0
  Lymphocytes >12*10^9 cells/L | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils ≤1.0*10^9 cells/L | 0 | 0 | 1 | 0 | 0 | 1
  Neutrophils <1.5*10^9 cells/L | 0 | 4 | 2 | 2 | 5 | 2
  Neutrophils ≥12*10^9 cells/L | 4 | 3 | 2 | 1 | 4 | 2
  RBC Count ≤3.3*10^12 cells/L | 0 | 0 | 0 | 0 | 0 | 0
  RBC Count ≥6.8*10^12 cells/L | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin ≤100 g/L | 1 | 5 | 3 | 3 | 3 | 3
  Platelet Count ≤100*10^9 cells/L | 0 | 0 | 0 | 0 | 0 | 1
  Platelet Count ≥600*10^9 cells/L | 0 | 2 | 1 | 0 | 1 | 0

11. Primary Outcome: Number of Participants With Abnormalities in Blood Chemistry Laboratory Data
Description: For each abnormality a subject can be counted once. If a subject has more than one occurrence of the same abnormality the highest toxicity grade is counted. ALT=alanine aminotransferase; AST=aspartate aminotransferase; ALP=alkaline phosphatase; GGT=gamma-glutamyl transferase; TSH=thyroid stimulating hormone, ULN=upper limit of normal.
Time Frame: Up to 72 Weeks
Population: Safety Population: all randomized participants who received study treatment; n=number of participants whose baseline value for 205MS202 (NCT00870740) was normal (i.e. not high or low) and who had at least one post-baseline value during the study.
Measure: Number; unit: participants
Arm/Group | Placebo + DAC HYP 150 mg | Placebo + DAC HYP 300 mg | DAC HYP 150 mg + Washout | DAC HYP 150 mg for 2 Years | DAC HYP 300 mg + Washout | DAC HYP 300 mg for 2 Years
Number analyzed (Participants) | 86 | 84 | 86 | 86 | 88 | 87
participants
  ALT ≤ULN; n=84,81,78,81,83,79 | 65 | 62 | 61 | 62 | 60 | 55
  ALT >1 to <3 ULN; n=84,81,78,81,83,79 | 18 | 17 | 16 | 19 | 20 | 20
  ALT 3 to 5 ULN; n=84,81,78,81,83,79 | 0 | 1 | 0 | 0 | 0 | 3
  ALT >5 to 10 ULN; n=84,81,78,81,83,79 | 1 | 1 | 1 | 0 | 2 | 0
  ALT >10 to 20 ULN; n=84,81,78,81,83,79 | 0 | 0 | 0 | 0 | 1 | 1
  ALT >20 ULN; n=84,81,78,81,83,79 | 0 | 0 | 0 | 0 | 0 | 0
  AST ≤ULN; n=85,81,81,84,85,84 | 72 | 66 | 71 | 63 | 68 | 62
  AST >1 to <3 ULN; n=85,81,81,84,85,84 | 13 | 14 | 9 | 20 | 14 | 18
  AST 3 to 5 ULN; n=85,81,81,84,85,84 | 0 | 1 | 1 | 1 | 2 | 2
  AST >5 to 10 ULN; n=85,81,81,84,85,84 | 0 | 0 | 0 | 0 | 0 | 2
  AST >10 to 20 ULN; n=85,81,81,84,85,84 | 0 | 0 | 0 | 0 | 0 | 0
  AST >20 ULN; n=85,81,81,84,85,84 | 0 | 0 | 0 | 0 | 1 | 0
  ALP ≤ULN; n=84,84,84,84,86,86 | 76 | 83 | 80 | 80 | 81 | 82
  ALP >1 to 2.5 ULN; n=84,84,84,84,86,86 | 8 | 1 | 4 | 4 | 5 | 4
  ALP >2.5 to 5 ULN; n=84,84,84,84,86,86 | 0 | 0 | 0 | 0 | 0 | 0
  ALP >5 to 20 ULN; n=84,84,84,84,86,86 | 0 | 0 | 0 | 0 | 0 | 0
  ALP >20 ULN; n=84,84,84,84,86,86 | 0 | 0 | 0 | 0 | 0 | 0
  GGT ≤ULN; n=81,79,81,82,84,82 | 74 | 71 | 74 | 74 | 73 | 73
  GGT >1 to 2.5 ULN; n=81,79,81,82,84,82 | 5 | 8 | 5 | 6 | 8 | 9
  GGT >2.5 to 5 ULN; n=81,79,81,82,84,82 | 2 | 0 | 2 | 2 | 2 | 0
  GGT >5 to 20 ULN; n=81,79,81,82,84,82 | 0 | 0 | 0 | 0 | 1 | 0
  GGT >20 ULN; n=81,79,81,82,84,82 | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin ≤ULN; n=81,79,83,81,85,80 | 74 | 73 | 81 | 76 | 78 | 75
  Total Bilirubin >1 to 1.5 ULN; n=81,79,83,81,85,80 | 5 | 6 | 2 | 4 | 4 | 5
  Total Bilirubin >1.5 to 3 ULN; n=81,79,83,81,85,80 | 2 | 0 | 0 | 1 | 2 | 0
  Total Bilirubin >3 to 10 ULN; n=81,79,83,81,85,80 | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin >10 ULN; n=81,79,83,81,85,80 | 0 | 0 | 0 | 0 | 1 | 0
  TSH-3rd Gen Abnormal; n=79,79,74,77,79,79 | 2 | 1 | 2 | 2 | 2 | 2
  Free Thyroxine (T4) Abnormal; n=78,80,73,73,80,79 | 4 | 4 | 5 | 4 | 4 | 3
  Total Thyroxine (T4) Abnormal; n=76,80,74,72,80,79 | 3 | 10 | 6 | 4 | 9 | 9

12. Primary Outcome: Number of Participants With Development of Anti-DAC Antibodies (ADAb) and Neutralizing Antibodies (NAb) Post-baseline
Description: Number of participants positive and negative for ADAb and NAb, based on all post-baseline immunogenicity assessments during treatment period and follow-up. Participants are stratified differently in this Outcome Measure as per the pre-specified statistical analysis plan.
Time Frame: Up to 72 weeks
Population: All participants in the Safety Population (all randomized participants who received study treatment) with a post-baseline ADAb assessment.
Measure: Number; unit: participants
Arm/Group | Placebo + DAC HYP | DAC HYP + Washout | DAC HYP for 2 Years
Number analyzed (Participants) | 169 | 171 | 170
participants
  ADAb Positive | 7 | 21 | 3
  ADAb Negative | 162 | 150 | 167
  NAb Positive | 4 | 4 | 1
  NAb Negative | 165 | 167 | 169

13. Secondary Outcome: Rate of Percentage Change From Baseline in Mean Total Brain Volume
Description: Total brain volume was measured by MRI and analyzed by a central reader. Rate of percentage change from baseline calculated using an analysis of covariance adjusting for baseline normalized brain volume. Baseline values = baseline for study 205MS202 (NCT00870740). Missing values post-baseline were imputed using the average value across subjects in the treatment group.
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: rate of percentage change
Groups:
- Placebo + DAC HYP 300 mg: Participants who previously received placebo in study received DAC HYP 300 mg SC injection every 4 weeks for a total of 13 doses.
Arm/Group | Placebo + DAC HYP 150 mg | Placebo + DAC HYP 300 mg | DAC HYP 150 mg + Washout | DAC HYP 150 mg for 2 Years | DAC HYP 300 mg + Washout | DAC HYP 300 mg for 2 Years
Number analyzed (Participants) | 79 | 76 | 61 | 64 | 63 | 62
rate of percentage change | -0.772 [-0.978 to -0.565] | -0.930 [-1.141 to -0.719] | -0.622 [-0.857 to -0.387] | -0.528 [-0.758 to -0.297] | -0.505 [-0.736 to -0.274] | -0.452 [-0.685 to -0.219]

ADVERSE EVENTS:
Time Frame: Study Entry Week 0 (Baseline; Week 52 Visit from study 205MS201 [NCT00390221]) through Week 72 ± 5 days or early termination.
Arm/Group | Placebo + DAC HYP 150 mg | Placebo + DAC HYP 300 mg | DAC HYP 150 mg + Washout | DAC HYP 150 mg for 2 Years | DAC HYP 300 mg + Washout | DAC HYP 300 mg for 2 Years
Serious Adverse Events (participants affected / at risk) | 15/86 | 11/84 | 18/86 | 15/86 | 14/88 | 11/87
Other Adverse Events (participants affected / at risk) | 43/86 | 37/84 | 47/86 | 38/86 | 45/88 | 43/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + DAC HYP 150 mg (N=86) | Placebo + DAC HYP 300 mg (N=84) | DAC HYP 150 mg + Washout (N=86) | DAC HYP 150 mg for 2 Years (N=86) | DAC HYP 300 mg + Washout (N=88) | DAC HYP 300 mg for 2 Years (N=87)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Basedow's disease (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chronic hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Meningitis aseptic (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Mycobacterium abscessus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis chronic (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Demyelination (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ischaemic neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Multiple sclerosis relapse (Nervous system disorders) | 9 | 7 | 12 | 9 | 12 | 5
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0
Mental disorder due to a general medical condition (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Glomerulonephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mesangioproliferative glomerulonephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Breast inflammation (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Pityriasis rubra pilaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + DAC HYP 150 mg (N=86) | Placebo + DAC HYP 300 mg (N=84) | DAC HYP 150 mg + Washout (N=86) | DAC HYP 150 mg for 2 Years (N=86) | DAC HYP 300 mg + Washout (N=88) | DAC HYP 300 mg for 2 Years (N=87)
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 1 | 5 | 2 | 1
Fatigue (General disorders) | 5 | 1 | 2 | 3 | 4 | 3
Pyrexia (General disorders) | 2 | 1 | 2 | 1 | 6 | 5
Nasopharyngitis (Infections and infestations) | 12 | 8 | 11 | 10 | 10 | 15
Oral herpes (Infections and infestations) | 5 | 1 | 6 | 1 | 6 | 2
Pharyngitis (Infections and infestations) | 5 | 3 | 4 | 5 | 2 | 5
Respiratory tract infection viral (Infections and infestations) | 3 | 3 | 5 | 1 | 4 | 2
Upper respiratory tract infection (Infections and infestations) | 6 | 4 | 7 | 9 | 6 | 7
Alanine aminotransferase increased (Investigations) | 2 | 2 | 3 | 4 | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 7 | 2 | 2 | 2 | 3
Headache (Nervous system disorders) | 5 | 4 | 5 | 4 | 8 | 6
Multiple sclerosis relapse (Nervous system disorders) | 16 | 13 | 25 | 13 | 17 | 13
Rash (Skin and subcutaneous tissue disorders) | 3 | 5 | 5 | 4 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.